CLINICAL TRIAL: NCT07075263
Title: Smoking Among Resident Physician and Their Role in Smoking Cessation Advice
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Lecturer faculty of medicine, Mansoura University Hospital
Other Study IDs: MS.21.05.1492
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
Keywords: Smoking; Smoking cessation; Resident physicians
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resident physicians: whole total resident physicians number at Mansoura university hospital in 2023
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A self-administered structured questionnaire

SUMMARY:
smoking is a key modifiable risk factor that greatly increases the likelihood of 2 dying young from cancer, heart disease, and lung disorders The World Health Organization (WHO) reports that 3 tobacco products are used by one-third of the world's population, and that 90% of tobacco users began using 4 them before the age of 18.

DETAILED DESCRIPTION:
The majority of smokers make multiple unsuccessful attempts to stop 5 smoking before attaining long-term abstinence, with over half of these attempts culminating in a relapse. 6 Healthcare professionals are essential in helping people stop smoking. According to professional guidelines and 7 the World Health Organization (WHO), doctors should actively encourage smokers to give up. Aim of this work 8 was to explore the knowledge, attitude and practice of resident physicians about smoking cessation program and 9 the effect of their smoking habits on smoking cessation advice for patients.

ELIGIBILITY:
Inclusion Criteria:

* whole total resident physicians number at Mansoura university hospital in 2023

Exclusion Criteria:

* refuse to share or had a vacation from work

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study included the whole total resident physicians number at Mansoura university hospital in 2023
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Smoking cessation awareness | 6 months
  questions which cover counseling or receiving of therapy for smoking cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AbdElmoniem, Principal Investigator — Lecturer of chest medicine faculty of medicine Mansoura university
Locations (1):
- Mohamed AbdElmoniem, Al Mansurah, Egypt